CLINICAL TRIAL: NCT05031663
Title: Effect of Daily Consumption of Almonds on Immune Strength and Response to Flu Vaccination in Overweight Middle -Aged Men: A Randomized Controlled Study
Brief Title: Effect of Almonds on Immune Strength and Response to Flu Vaccination in Overweight Older Men and Postmenopausal Women: A Randomized Controlled Study
Acronym: Almond Immune
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Joan Sabate,DrPH, MD, Professor of Nutrition, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5210259
Record Dates: First submitted 2021-07-06; First posted 2021-09-02 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Immune Response; Inflammation
Keywords: Almonds; Immunity; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: this will be a parallel, free-living, randomized controlled trial, where 66 middle-aged men and post menopausal women will be randomized to receive either the almonds or control
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and outcome assessor will not be aware which participant is in what arm. The participant and the care provider will know about the treatment allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almonds (Experimental): The almond group will receive 15% of their daily energy intake in the form of almonds
  Interventions: Dietary Supplement: Almond group
- Control (Placebo Comparator): The control group will be encouraged to continue their usual diet but completely avoid almonds and restrict other nuts to less than 2 servings per week
  Interventions: Dietary Supplement: Control Group

INTERVENTIONS:
Dietary Supplement: Almond group — Participants in the Almond group will receive 15% of their daily energy intake in the form of almonds as a snack
  Arms: Almonds
Dietary Supplement: Control Group — The control group will continue their usual diet but will completely avoid almonds and restrict other nuts to less than 2 servings per week
  Arms: Control

SUMMARY:
This research study will test the effects of almonds on immune functions and immune response to influenza vaccine in overweight middle-aged men and postmenopausal women

DETAILED DESCRIPTION:
The proposed study is a parallel-group, free-living, observer-blind, randomized controlled dietary intervention trial on 66 overweight middle-aged men and post menopausal women. This study will be carried out in two phases: Phase 1 will examine the effects of almonds on clinically relevant markers of immune function, and Phase 2 will assess the antibody response to influenza vaccination following almond consumption. Participants will attend a baseline clinic and will be randomized to one of two groups. The Almond group will receive 15% of daily energy intake in the form of almonds as a snack and the Control group will continue thier usual diet but completely avoid almonds and restrict other nuts to less than 2 servings per week. The intervention will be for 12 weeks, at which time both group participants will receive the influenza vaccination, and continue the same dietary intervention for another 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Overweight men and post menopausal women (Basal Metabolic Index 25-32)
* Age limit between 40-70 years
* Be able to commute to Loma Linda University

Exclusion Criteria:

* Intolerance or allergy to almonds
* Bad dentures, inability to chew almonds
* Regular intake of almonds and or other nuts
* Use of immune boosting supplements
* Exposure to antibiotics and corticosteroids immediately prior to study
* Have received influenza vaccination in past 10 months
* Uncontrolled chronic disease and psychiatric illness

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
changes in lymphocyte populations | baseline to 12 weeks
  Immunophenotyping will be performed by flow cytometry to measure the number of T helper, T cytotoxic, Naïve and memory cells and B cells
changes in lymphocyte activity and cytokine production | baseline to 12 weeks
  PBMC cells will be separated from blood, activated and cultured using phytohemagglutinin (PHA). Inflammatory cytokine production will be measured in the resulting supernatant using ELISA
changes in natural killer (NK) cell activity | baseline to 12 weeks
  The NK degranulation assay will be performed on blood samples. The test will be conducted using a modified flow cytometry method that measures the expression of CD107a
changes in serum inflammatory cytokine concentration | baseline to 12 weeks
  Changes in the concentrations of the inflammatory cytokines will be performed on serum using enzyme-linked immunoassay (ELISA)
changes in complete blood count (CBC) | baseline to 12 weeks
  changes in the complete blood count will be performed on whole blood with the use of an automated hematology analyzer at a certified clinical facility

SECONDARY OUTCOMES:
changes in upper respiratory infection questionnaire score | baseline to 28 weeks
  Upper respiratory tract infections will be tracked using the Jackson and Dowling questionnaire. The questionnaire will be completed daily by participants, either manually or electronically , throughout the 28-week study period. The scale for the questionnaire is from 0-42. The higher score means worse outcome.
changes in blood zinc levels | baseline to 12 weeks
  Zinc levels in blood will be analyzed in trace element- free tubes and assayed by atomic absorption spectrophotometry using standard reference material obtained from the National Institute of Standards and Technology to check the accuracy and precision of the determinations

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabate, DrPh, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University School of Public Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No